CLINICAL TRIAL: NCT01892592
Title: Discovering Healthcare Innovations to Address Disparities in Stroke
Brief Title: Discovering Healthcare Innovations to Address Disparities in Stroke (DIADS)
Acronym: DIADS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Kaiser Permanente (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CN-12SSidn-06-H
Record Dates: First submitted 2013-03-21; First posted 2013-07-04 (Estimated); Last update posted 2022-05-20 (Actual); Status verified 2022-05

CONDITIONS: Hypertension
Keywords: Hypertension; African American; Health Disparities; Stroke; Cardiovascular Disease
MeSH Terms: conditions — Hypertension; Stroke; Cardiovascular Diseases | interventions — Diet; Behavior Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Usual Care (No Intervention): No Interventions
- Medication enhancement (No Intervention): Pharmacist will optimize current Kaiser medication protocol for treatment of hypertension.
- Diet and Lifestyle Arm (Experimental): Patients will receive up to 16 wellness coaching sessions focusing on DASH doest and lifestyle changes - Behavioral Intervention
  Interventions: Behavioral: Diet and Lifestyle

INTERVENTIONS:
Behavioral: Diet and Lifestyle — Patients will receive up to 16 phone based coaching sessions
  Other Names: Behavioral Interventions; Wellenss Coaching
  Arms: Diet and Lifestyle Arm

SUMMARY:
The goal of this pragmatic study is to improve hypertension (HTN) control rate in blacks and to reduce racial disparity in HTN control. To accomplish this, the investigators propose to perform a cluster randomized controlled trial at the primary care provider (PCP) level and including 191 PCPs within KPNC East Bay Service Area with more than 45,000 patients in the HTN registry of which approximately 15,000 are black. The investigators will randomize all PCP patient panels to a three-arm trial to receiving either 1) usual care; or 2) culturally tailored diet and lifestyle coaching; or 3) an intensified BP management protocol with pharmacotherapy. The "Shake, Rattle and Roll" trial is named for: 1) "shake" the salt habit; 2) "rattle" the intensity of current BP management; and 3) design the interventions with the goal of being able to adapt and "roll" them out to community clinics outside of a managed care system. Primary research question: whether a primary prevention intervention of either diet and lifestyle coaching or an intensive pharmacotherapy protocol is more effective than usual care in improving rates of HTN control in blacks and thereby reducing disparities between black and white. Primary aim: By implementing either intervention, the investigators will reduce the disparity in hypertension control rates between blacks and whites by 4% at 1 year post-study enrollment. Hypothesis: Among blacks with HTN, a diet/lifestyle coaching intervention or an intensified BP management protocol will result in an increase in HTN control rate compared to usual care. Primary outcome: the proportion of patients with sustained BP control at 1 year post-study enrollment.

DETAILED DESCRIPTION:
Kaiser Permanente Northern California (KPNC) serves a population of over 3 million enrollees, representative of the socio-demographic characteristics of the San Francisco Bay Area, Santa Rosa, and Sacramento except for under-representation of the very rich and very poor.78 KPNC is the largest nonprofit integrated health care organization in the country, with 22 hospitals and 44 outpatient facilities, and cares for 30% of the population in the region. The majority of Californians are managed in four large hospital networks, so the KPNC system is a model for the 167 Program Director/Principal Investigator (Last, First, Middle): Sidney, Stephen, MD, MPH PHS 398/2590 (Rev. 06/09) Page Continuation Format Page prevalent system of care in the state. An effective system-wide intervention in KPNC would likely be generalizable and feasible in the other healthcare networks in the State and, thus, could benefit the population more broadly. The project focuses on the East Bay Service Area (EBSA) because approximately one-third of African American KPNC members with HTN receive care within this geographical area. The East Bay area, home of the flagship Oakland Medical Center and Richmond Medical Center, comprises 12 cities and municipalities within the Alameda County and the western section of Contra Costa County. From Kaiser Permanente's inception in 1945, the nonprofit organization has led with innovation, beginning with its prepaid health care services offered to Richmond shipyard workers during World War II. Today, the Richmond and Oakland Medical Centers are home to about 700 physicians and 5,600 employees who serve over a quarter of a million members yearly.

Kaiser Permanente East Bay has expanded its services for West Contra Costa members. The brand new Pinole Medical Office Building, just eight miles from the Richmond Medical Center offers convenient access to members in the East Bay Area, which includes Pinole, El Sobrante, Hercules, Rodeo and Crockett.

The Pinole center provides adult medicine, family practice, pediatrics, obstetrics/gynecology, radiology, a lab, a pharmacy, and health education. For emergency services, members go to the Richmond Medical Center, and for labor and delivery services, the Oakland Medical Center. The fourth member of the EBSA is the Alameda Medical Center which offers services for internal medicine, gynecology, pediatrics, pharmacy, and members outreach. Using KPNC as a model offers several major advantages. Members generally remain in the plan for many years, with 94% retention at 1 year and 84% retention at 5 years among enrollees 65-74 years old.

Sources of electronic medical data are extensive and easy to manipulate. They will be combined to produce an electronic registry of patients with uncontrolled HTN (Figure - Electronic Registry; source of data provided in brackets). The following information is available from electronic medical record (EMR) system:

* Inpatient discharge abstracts with primary and secondary diagnoses and procedures coded by a trained medical records analyst.
* Inpatient discharge abstracts for all out-of-plan hospital admissions.
* Emergency-department and outpatient diagnoses coded by the treating physician.
* All outpatient records including BP measurements.
* All radiology reports generated by reviewing radiologists.
* Listing of all major health problems generated and frequently updated by all treating physicians.
* Cardiologist interpretations of all ECGs.
* Reports from all clinical laboratory studies.
* Listing of all outpatient filled prescriptions and completed inpatient medication orders.

The EMR databases have been validated extensively and, in combination, have been shown to accurately reflect a number of disease diagnosis, comorbidities, and outcomes.79-81 The KPNC Division of Research maintains a mortality database for all KPNC members dating back to 1971. The primary sources of mortality data are the California Department of Health Services, which maintains a registry of deaths and their causes, and Social Security mortality files for more recent deaths. With the recent loss of the utility of the Social Security mortality files, we have made arrangements to have more frequent updates (quarterly or semi-annually) from the California Department of Health Services so that our mortality file will be current until the approximately past 6 months. Mortality will also be assessed from the KPNC EMR if they occur during a hospitalization. The "Shake, Rattle and Roll" trial is named for: 1) "shake" the salt habit; 2) "rattle" the intensity of the current clinical BP protocol; and 3) design the interventions with the ultimate goal of being able to adapt and "roll" out the interventions to community clinics outside of the managed care system.

Randomization There are 194 PCPs in the EBSA with 191 providers having African Americans in their patient panels.

The unit of randomization will be the primary care providers in the EBSA (N=191) who have black patients in their panels. The other 3 PCPs can be randomized into the study at a later date if and when they add African American patients to their panels. All PCPs will be randomized to one of the 3 arms. To the extent possible, we will strive to have an approximately equal number of African Americans with HTN in each arm of the trial (approximately 1896 with uncontrolled HTN expected per group). This will be accomplished by using stratified black patients with hypertension in each clinician's panel.

With the intensified BP protocol intervention, because it is a quality improvement effort, randomizing at the provider level will allow all African American patients with HTN to be targeted for the intervention should their BP ever become uncontrolled. We will not need to ask patients if they are willing to participate given the intervention is an extension of the usual care model with more intensive focus on aggressive HTN management for African Americans. We will seek a waiver of informed consent for the intervention from our local Institutional Review Board (IRB) and have been advised by the IRB administrator that the waiver will likely be approved by the IRB.

Being able to include all African Americans in this intervention will increase the generalizability of the study findings. With the diet and lifestyle coaching intervention, randomizing at the provider level will also allow us to invite all African American patients with uncontrolled HTN to participate in this intervention. Even though the materials used in developing this intervention are available within KPNC, a formal coaching program for diet and lifestyle effects on HTN is currently non-existent. We will send out letters to inform eligible patients of this on-going improvement project. The patients will have the option of opting out of the study by returning a stamped envelope to us. If the patients choose not to opt out, then a research staff will contact them to discuss enrollment as scheduled (Figure - study diagram, above). As detailed in the Statistical Analysis Section we anticipate enrollment of approximately 1896 blacks with uncontrolled HTN to each arm of the study spread out over a 2-year period. The randomization process of all PCPs will be carried out by a programmer at the KPNC DOR offices (Oakland, CA).

ELIGIBILITY:
Inclusion Criteria:

* African American
* > age 18
* Blood Pressure >140/90

Exclusion Criteria:

-

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 1761 (Actual)
Dates: Start 2013-06; Primary Completion 2015-06 (Actual); Study Completion 2018-06 (Actual)

PRIMARY OUTCOMES:
Percentage of Blacks / African Americans with HTY with controlled blood pressure (BP) after 1 year. | 1 year
  Percentage of Blacks / African Americans with HTY with controlled blood pressure (BP) after 1 year.

CONTACTS AND LOCATIONS:
Overall Officials: Mai N Nguyen-Huynh, MD, Principal Investigator — Research Scientist
Locations (1):
- Kaiser Permanene Oakland Medical Center, Oakland, California, United States

REFERENCES:
- [Derived] Nguyen-Huynh MN, Young JD, Ovbiagele B, Alexander JG, Alexeeff S, Lee C, Blick N, Caan BJ, Go AS, Sidney S. Effect of Lifestyle Coaching or Enhanced Pharmacotherapy on Blood Pressure Control Among Black Adults With Persistent Uncontrolled Hypertension: A Cluster Randomized Clinical Trial. JAMA Netw Open. 2022 May 2;5(5):e2212397. doi: 10.1001/jamanetworkopen.2022.12397. PMID 35583869
- [Derived] Nguyen-Huynh MN, Young JD, Alexeeff S, Hatfield MK, Sidney S. Shake Rattle & Roll - Design and rationale for a pragmatic trial to improve blood pressure control among blacks with persistent hypertension. Contemp Clin Trials. 2019 Jan;76:85-92. doi: 10.1016/j.cct.2018.11.012. Epub 2018 Nov 28. PMID 30500558